CLINICAL TRIAL: NCT01307293
Title: Randomized Controlled Trial of a Brief Cognitive Behavioral Intervention Designed to Prevent and Reduce Symptoms of Posttraumatic Stress in Mothers of Preterm Infants.
Brief Title: Prevention of Postpartum Traumatic Stress (PTSD) in Mothers With Preterm Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-02172011-7504
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): 6-12 sessions of Cognitive Behavior Therapy to address PTSD symptoms and parenting issues related to premature infants.
  Interventions: Behavioral: Cognitive behavior therapy
- Placebo comparison (No Intervention): Education regarding NICU parenting issues.

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — 6 or 12 sessions of cognitive behavior therapy.
  Arms: Cognitive Behavior Therapy

SUMMARY:
The purpose of the study includes:

1. To develop a treatment manual and pilot test this treatment intervention which is designed to prevent and reduce psychological distress in parents who have infants hospitalized in the neonatal intensive care unit (NICU).
2. To conduct a treatment intervention study in which parents of NICU infants will receive a 6-12 session treatment designed to reduce psychological distress, and to compare outcomes with parents who do not receive the intervention.

We hope to learn whether or not a simple psychotherapeutic and psychoeducational intervention offered to parents of NICU infants can prevent or minimize the development of symptoms of psychological distress in parents, including symptoms of anxiety and depression and posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
There are three phases to this research study:

1. DEVELOPMENT OF A TREATMENT MANUAL TO HELP REDUCE PSYCHOLOGICAL DISTRESS IN PARENTS OF NICU INFANTS.

   We currently have pilot data on a three session intervention designed to reduce psychological distress in NICU parents. In this phase of hte study, we plan to augment this intervention by adding an additional three sessions for a total of six sessions which will comprise our new treatment manual. To accomplish this, we will conduct a comprehensive review of the content of all current empirically based cognitive behavior therapy (CBT) treatments for PTSD, abstract the key elements, compare the key elements with our current treatment for PTSD and construct a fourth session using a combination of Stress Inoculation Training techniques (including relaxation training, thought stopping, cognitive restructuring) and imaginal re-exposure. A similar process will be used to identify parent-child interventions currently available used with premature or other vulnerable young children. The redefinition of the infant and reeducation of the mother to promote sensitivity toward and attachment with the infant are likely topics.
2. PILOT THE MANUALIZED TREATMENT IN AN OPEN TRIAL WITH 10 NICU MOTHERS, SOLICIT FEEDBACK AND MODIFY INTERVENTION SESSIONS.

   To obtain clinically relevant feedback and prepare for any unforeseen logistical issues, we will pilot the six session treatment intervention in 10 mothers whose newborns are hospitalized in the LPCH NICU. The recruited parents will be representative of the population of mothers that the intervention is intended for-English and Spanish speaking mothers of infants >= 28 weeks, over 1000 grams, born at LPCH or transferred within 72 hours with CRIB scores, a measure of medical severity, of 15 or less. Children transferred for cardiac surgery and those with congenital abnormalities will not be eligible. Mothers will be approached by a member of the NICU staff within 72 hours of the infant's admission to the NICU. The mother will be given an information sheet about the project and invited to speak with the study coordinator. Potential subjects who give informed consent will complete the three screening instruments, the Stanford Acute Stress Reaction Questionnaire (SASRQ), Beck Anxiety Inventory (BAI) and Beck Depression Inventory-I (BDI I) and the sociodemographic questions.

   Within 48 hours, one of the study psychologists, will contact enrolled mothers, establish a schedule for the 6 sessions and initiate the course of treatment. The sessions will be individual and held at a time and location convenient for the mother. We expect that most sessions will be in the LPCH NICU in private offices suitable for therapy sessions. Should the infant be discharged from the NICU prior to the 6th session, the remaining sessions will be scheduled at home, LPCH or the Department of Psychiatry. Following the 6th session, the mothers will be contacted by the study coordinator who will administer the instruments chosen for the post intervention assessment and assess satisfaction with the treatment sessions. Specific questions will include: What did you like/dislike about the treatment?; Which sessions were most/least helpful?; Could the treatment be structured differently?; Was the timing/length of the sessions appropriate?; Were the techniques taught useful?; How satisfied were you with this intervention? All evaluation materials including changes in pre/post scores on our instruments will be summarized and presented to our Scientific Advisory Group. Once consensus is reached on the revised manual, the manual will be rewritten to incorporate feedback and data obtained in the pilot study.
3. CONDUCT A RANDOMIZED TRIAL OF THE TREATMENT INTERVENTION COMPARED TO AN INFORMATION, USUAL CARE, SUPPORT CONTROL CONDITION.

Eligible mothers (N=100) will be randomly assigned to receive either: (1) the manual driven, CBT-based trauma focused plus mother redefinition/education intervention; or (2) information, usual care/support. The intervention is expected to last 3 weeks with two 45-55 minute sessions weekly. Participants in both conditions will be assessed at baseline, within one week after the completion of the intervention or at 4-5 weeks for the control group and at 6-months post-baseline.

The information/usual-care/support condition was chosen to control for possible symptom changes due to routine clinical contacts common in the NICU, the effect of time, the effect of attention and any effects due to repeated assessments. Parents in the information/usual care/support group will receive one 45 minute information session on the policy, procedures and environment of the NICU by a Neonatal Nurse Practitioner (Table 4). We have chosen to use a Nurse Practitioner for the information comparison because this is a role they often assume at LPCH. This session is based on an LPCH Hospital Information Packet that is routinely distributed to all NICU parents, although generally without any instruction or face-to-face review of its content. Women in this group will be followed up by telephone or in the NICU one week after the information session to answer any questions that they may have. In addition, mothers will be referred to the existing parent mentor program for support and coping strategies. By adding the parent mentor support we expect that the contact will be similar to the intervention group and, thus, will approximate an attention-matched comparison condition. Mothers in this group will also receive the care that is typical for NICU parents including contacts with nurses, physicians, social workers, chaplaincy and developmental psychologists.

Thirty of the participants in the intervention arm will be randomized to receive an expanded intervention of 6 additional sessions (sessions 7-12). These sessions will elaborate on the themes identified in Session 4 and follow the current models of PTSD treatment that generally provide a minimum of 12 sessions. These sessions will likely use cognitive restructuring to address distortions about the NICU experience. Specific issues explored will be individualized to each parent but may include parental guilt, parental anxiety about their infant's medical health, and difficulties related to the perceived absence of a parental role. There will also be a strong emphasis on the use of stress inoculation training to assist parents in developing strategies to manage trauma symptoms. The 30 participants in the intervention arm who are not randomized to the expanded intervention will be offered contact with the existing parent mentor program. Parent mentors offer support, coping strategies and suggestions on how to normalize life after the NICU hospitalization. Should an infant die, the mother will be disenrolled from the study and assisted with a referral for conventional mental health support services.

ELIGIBILITY:
Inclusion Criteria:

English and Spanish-speaking mothers greater than 18 years of age of infants in the LPCH NICU >=26 weeks of gestation are eligible for screening.

Exclusion Criteria:

1. Mothers of children awaiting cardiac surgery, those who have congenital abnormities and those who are unlikely to survive, will be excluded.
2. Mothers of NICU infants who are found on their routine clinical psychosocial evaluation to be at high psychiatric risk (i.e., those with either psychotic symptoms or suicidal or infanticidal ideation) will also be excluded. These parents, however, will be referred for and receive appropriate mental health intervention.
3. Mothers who do not speak English or Spanish, or who do not have the ability to understand the questionnaires will be excluded.
4. Mothers who have active and current symptoms of suicidal ideation, or psychotic symptoms (delusions or hallucinations) as identified by self report or following a diagnostic interview will be excluded from the study, but will also be referred for emergency psychiatric evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Davidson Trauma Scale | 6 months
BDI-II | 6 months

SECONDARY OUTCOMES:
CAPUTE | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Shaw, Principal Investigator — Stanford University; Sarah McCue Horwitz, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Shaw RJ, St John N, Lilo E, Jo B, Benitz W, Stevenson DK, Horwitz SM. Prevention of traumatic stress in mothers of preterms: 6-month outcomes. Pediatrics. 2014 Aug;134(2):e481-8. doi: 10.1542/peds.2014-0529. PMID 25049338
- [Result] Shaw RJ, St John N, Lilo EA, Jo B, Benitz W, Stevenson DK, Horwitz SM. Prevention of traumatic stress in mothers with preterm infants: a randomized controlled trial. Pediatrics. 2013 Oct;132(4):e886-94. doi: 10.1542/peds.2013-1331. Epub 2013 Sep 2. PMID 23999956
- [Derived] Horwitz SM, Storfer-Isser A, Kerker BD, Lilo E, Leibovitz A, St John N, Shaw RJ. A model for the development of mothers' perceived vulnerability of preterm infants. J Dev Behav Pediatr. 2015 Jun;36(5):371-80. doi: 10.1097/DBP.0000000000000173. PMID 25961903